CLINICAL TRIAL: NCT04722536
Title: Effectiveness of CERvico-isthmic CErclage in Increasing the Rate of Live Births in Case of a History of Late Miscarriage and/or Premature Delivery
Brief Title: Effectiveness of Cervico-isthmic Cerclage
Acronym: CERCEI LB
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1088; 2020-A03187-32 (Other: ID-RCB)
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Cerclage, Cervical; Cervical Insufficiency
Keywords: cervico-isthmic cerclage; cerclage; cervico-isthmic; cervical insufficiency; miscarriage; prematurity
MeSH Terms: conditions — Uterine Cervical Incompetence; Abortion, Spontaneous; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervico-isthmic cerclage: Are included in this group the women who underwent cervico-isthmic cerclage between January 1, 2010 and April 1, 2019, in 3 hospitals of the Hospices Civils de Lyon, respecting the inclusion and exclusion criteria, to assess the primary and secondary outcomes before and after performing the cerclage.
  Interventions: Procedure: Cervico-isthmic cerclage

INTERVENTIONS:
Procedure: Cervico-isthmic cerclage — There is no intervention in this study. It's an observational retrospective study, before/after.

SUMMARY:
This study compares the rate of live births before and after cervico-isthmic cerclage in 3 hospitals in the last 10 years. The hypothesis is that cerclage significantly increases the rate of live births in women with cervical insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* History of premature delivery or late miscarriage unrelated to maternal pathology, chorioamnionitis, fetal or placental pathology
* Patient aged over 18 at the time of the phone call
* Cerclage performed according to the Benson technique verified on the operative report
* Cerclage performed in one of the 3 obstetric gynecology departments of the CHU de Lyon (Lyon Sud, Croix Rousse and HFME) between January 1, 2010 and April 1, 2019

Exclusion Criteria:

* History of trachelectomy
* Surgical technique not specified or not deductible from the operating report
* Refusal to participate in the study
* Patient under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had cervico-isthmic cerclage between January 1, 2010 and April 1, 2019, in 3 University Hospitals of Lyon (Lyon Sud Hospital, HFME Hospital and Croix-Rousse Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-06-13 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Number of live birth ≥ 24 weeks of gestation or before 24 weeks of gestation with active neonatal intensive care, among pregnancies progressing after 14 weeks of gestation. | Day 0 (At Inclusion)
  We collect the data necessary to assess the outcomes in the medical charts. When data is missing, we will call patients (telephone interview) and ask them a few questions related to their gynecological and obstetric history.

CONTACTS AND LOCATIONS:
Overall Officials: DEBORAH GAVANIER, MD, Principal Investigator — Service de gynécologie-obstétrique - Centre Hospitalier Lyon Sud
Locations (3):
- France (3):
  - Hôpital Femme Mère Enfant (HFME) - Hospices Civils de Lyon, Bron
  - Hôpital de la Croix Rousse - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Lyon Sud (CHLS) - Hospices Civils de Lyon, Pierre-Bénite